CLINICAL TRIAL: NCT06228703
Title: The Effects of Different Flow Settings on Lung Impedance Using Two New HFNC Devices: A Randomized Crossover Study on Healthy Volunteers
Brief Title: The Effects of Different Flow Settings on Lung Impedance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HFNC-05
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: high-flow nasal cannula; ventilation distribution; lung impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Airvo 3 high-flow nasal cannula device with flow set at 20 L/min (No Intervention): A new high-flow nasal cannula device (Airvo 3) will be used in the study, with the flow set at 20 L/min
- HFT 750 high-flow nasal cannula device with flow set at 20 L/min (No Intervention): A new high-flow nasal cannula device (HFT 750) will be used in the study, with the flow set at 20 L/min
- Airvo 3 high-flow nasal cannula device with flow set at 40 L/min (Experimental): Airvo 3 will be used with the flow set at 40 L/min
  Interventions: Device: High-flow nasal cannula device with flow setting at 40 L/min or higher
- Airvo 3 high-flow nasal cannula device with flow set at 60 L/min (Experimental): Airvo 3 will be used with the flow set at 60 L/min
  Interventions: Device: High-flow nasal cannula device with flow setting at 40 L/min or higher
- HFT 750 high-flow nasal cannula device with flow set at 40 L/min (Experimental): HFT 750 will be used with the flow set at 40 L/min
  Interventions: Device: High-flow nasal cannula device with flow setting at 40 L/min or higher
- HFT 750 high-flow nasal cannula device with flow set at 60 L/min (Experimental): HFT 750 will be used with the flow set at 60 L/min
  Interventions: Device: High-flow nasal cannula device with flow setting at 40 L/min or higher

INTERVENTIONS:
Device: High-flow nasal cannula device with flow setting at 40 L/min or higher — Eligible participants will use the high-flow nasal cannula device (Airvo3 or HFT 750) with flow set at 40 L/min or higher
  Other Names: HFNC flow at 40 L/min or higher
  Arms: Airvo 3 high-flow nasal cannula device with flow set at 40 L/min; Airvo 3 high-flow nasal cannula device with flow set at 60 L/min; HFT 750 high-flow nasal cannula device with flow set at 40 L/min; HFT 750 high-flow nasal cannula device with flow set at 60 L/min

SUMMARY:
This prospective, randomized crossover trial will enroll adult healthy volunteers. Initially, the subject's peak inspiratory flow will be measured using a mask connected with a respiratory monitor. Subsequently, the volunteers will undergo HFNC treatment at different flow settings while their peak inspiratory flow will be continuously monitored. The primary outcome of this study is the lung aeration with different flow settings. Secondary outcomes include the lung aeration with different devices, subject's comfort at different flow settings, and the correlation between the subject's peak inspiratory flow measured by HFNC and by a mask connected with a respiratory monitor.

DETAILED DESCRIPTION:
Background: High-flow nasal cannula (HFNC) is a device that can reduce the work of breathing (WOB) and improve oxygenation by providing a flow that matches or exceeds patient's peak inspiratory flow during tidal breathing. Despite its widespread use, there remains a lack of consensus regarding the optimal flow settings. Two new HFNC devices that can provide information regarding patient's peak tidal inspiratory flow breath by breath are recently available, which might help guide set and titrate the flow settings. This study aims to investigate the effects of different flow settings on lung impedance in a cohort of healthy volunteers by using the two new HFNC devices.

Methods: This prospective, randomized crossover trial will enroll adult healthy volunteers. Initially, the subject's peak inspiratory flow will be measured using a mask connected with a respiratory monitor. Subsequently, the volunteers will undergo HFNC treatment at different flow settings while their peak inspiratory flow will be continuously monitored. The primary outcome of this study is the lung aeration with different flow settings. Secondary outcomes include the lung aeration with different devices, subject's comfort at different flow settings, and the correlation between the subject's peak inspiratory flow measured by HFNC and by a mask connected with a respiratory monitor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 21-65 years old

Exclusion Criteria:

* Chronic pulmonary diseases, including COPD, interstitial lung disease, cystic fibrosis, etc.
* Uncontrolled asthma;
* Pregnancy
* Subjects who have cold/flu symptoms (sore throat, runny nose, fever, chills, coughing)
* Nose abnormalities that can affect the functionality of the nasal prongs

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JIE LI, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University, Forest Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] McKinstry S, Pilcher J, Bardsley G, Berry J, Van de Hei S, Braithwaite I, Fingleton J, Weatherall M, Beasley R. Nasal high flow therapy and PtCO2 in stable COPD: A randomized controlled cross-over trial. Respirology. 2018 Apr;23(4):378-384. doi: 10.1111/resp.13185. Epub 2017 Sep 22. PMID 28940962
- [Background] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Background] Li J, Albuainain FA, Tan W, Scott JB, Roca O, Mauri T. The effects of flow settings during high-flow nasal cannula support for adult subjects: a systematic review. Crit Care. 2023 Feb 28;27(1):78. doi: 10.1186/s13054-023-04361-5. PMID 36855198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult healthy volunteers were recruited at a single academic medical center through posted study invitations and direct approach. Individuals expressing interest were screened for eligibility, and those who met inclusion criteria provided written informed consent prior to participation
Pre-assignment Details: Adult healthy volunteers were recruited at a single academic medical center through posted study invitations and direct approach. Individuals expressing interest were screened for eligibility, and those who met inclusion criteria provided written informed consent prior to participation
Groups:
- Total Study Population: This randomized crossover study evaluated two high-flow nasal cannula devices. All 26 participants completed the three prespecified flow-setting conditions for each device in a randomized sequence.
Period: Device A - Flow Setting 1
Arm/Group | Total Study Population
Started | 26
Completed | 26
Not Completed | 0
Period: Device A - Flow Setting 2
Arm/Group | Total Study Population
Started | 26
Completed | 26
Not Completed | 0
Period: Device A - Flow Setting 3
Arm/Group | Total Study Population
Started | 26
Completed | 26
Not Completed | 0
Period: Device B - Flow Setting 1
Arm/Group | Total Study Population
Started | 26
Completed | 26
Not Completed | 0
Period: Device B - Flow Setting 2
Arm/Group | Total Study Population
Started | 26
Completed | 26
Not Completed | 0
Period: Device B - Flow Setting 3
Arm/Group | Total Study Population
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Study Population: This randomized crossover study assigned all participants to receive each of the study treatments in a randomized order. All 26 participants contributed baseline demographic data to this single group.
Arm/Group | Total Study Population
Number analyzed (Participants) | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years] — age
  years | 27 [25 to 38]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All enrolled participants (n=26) were included in this baseline analysis.
  Participants
    Female | 18
    Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — This table reports participant self-identified race and ethnicity categories as collected during the study Population: All enrolled participants (n=26) were included in this baseline analysis.
  Participants
    Caucasian | 11
    Asian | 6
    Hispanic/Latino | 6
    African American | 2
    Other | 1
Height [Median (Inter-Quartile Range); unit: centimeter] — Population: All enrolled participants (n=26) were included in this baseline analysis.
  centimeter | 163 [157 to 170]
weight [Median (Inter-Quartile Range); unit: kilogram] | 68.0 [59.8 to 83.8]

OUTCOME MEASURES:

1. Primary Outcome: Change in End-expiratory Lung Impedance From Baseline Measured by Electrical Impedance Tomography (EIT)
Description: End-expiratory lung impedance (EELI) was measured continuously using electrical impedance tomography (EIT). For each flow-setting condition, EELI values were averaged over a stable 1-minute period. The outcome represents the change in EELI (in arbitrary impedance units) from each participant's baseline measurement prior to intervention. Positive values indicate an increase in end-expiratory lung volume compared to baseline, while negative values indicate a decrease. EIT impedance units are dimensionless and device-specific and are used to represent relative changes in ventilation and lung volume.
Time Frame: Up to 4 hours
Population: All enrolled participants (n=26) were included in this baseline analysis.
Measure: Mean (Standard Deviation); unit: Change in EELI (arbitrary units)
Arm/Group | Total Study Population
Number analyzed (Participants) | 26
Change in EELI (arbitrary units)
  EELI change with HFNC 20 L/min compared to baseline for HFT device | 9 (44)
  EELI change with HFNC 40 L/min compared to baseline for HFT device | 74 (80)
  EELI change with HFNC 60 L/min compared to baseline for HFT device | 132 (104)
  EELI change with HFNC 20 L/min compared to baseline for AIRVO device | 7 (44)
  EELI change with HFNC 40 L/min compared to baseline for AIRVO device | 71 (71)
  change with HFNC 60 L/min compared to baseline for AIRVO device | 111 (77)

2. Secondary Outcome: Changes in Respiratory Rates Compared to Baseline
Description: Respiratory rate was measured as breaths per minute. Change was calculated as the value during each HFNC flow condition minus the baseline respiratory rate. Positive values indicate an increase in respiratory rate, and negative values indicate a decrease.
Time Frame: Up to 4 hours
Population: All enrolled participants (n=26) were included in this baseline analysis.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Total Study Population
Number analyzed (Participants) | 26
breaths per minute
  Changes in respiratory rates at HFNC 20 L/min compared to baseline for HFT device | -1.6 (3.0)
  Changes in respiratory rates at HFNC 40 L/min compared to baseline for HFT device | -3.7 (5.6)
  Changes in respiratory rates at HFNC 60 L/min compared to baseline for HFT device | -5.0 (4.2)
  Changes in respiratory rates at HFNC 20 L/min compared to baseline for AIRVO device | -3.1 (3.2)
  Changes in respiratory rates at HFNC 40 L/min compared to baseline for AIRVO device | -3.1 (4.0)
  Changes in respiratory rates at HFNC 60 L/min compared to baseline for AIRVO device | -4.8 (6.1)

3. Secondary Outcome: Subject's Comfort Level
Description: Comfort level reported by participants using a visual numerical scale ranging between 0 (extreme discomfort) and 10 (very comfortable) at the end of each flow setting
Time Frame: Up to 4 hours
Population: All enrolled participants (n=26) were included in this baseline analysis.
Measure: Median (Inter-Quartile Range); unit: Score (0-10)
Arm/Group | Total Study Population
Number analyzed (Participants) | 26
Score (0-10)
  Comfort level at HFNC 20 L/min for HFT device | 9 [9 to 10]
  Comfort level at HFNC 40 L/min for HFT device | 8 [7 to 8]
  Comfort level at HFNC 60 L/min for HFT device | 7 [6 to 8]
  Comfort level at HFNC 20 L/min for AIRVO device | 9 [9 to 9]
  Comfort level at HFNC 40 L/min for AIRVO device | 8 [8 to 9]
  Comfort level at HFNC 60 L/min for AIRVO device | 8 [7 to 8]

ADVERSE EVENTS:
Time Frame: From the start of the experimental session until completion of all flow conditions (up to 4 hours)
Description: Adverse events were monitored throughout the experimental session by direct observation. The study involved healthy volunteers undergoing brief respiratory interventions, with no clinical treatments or follow-up. No differences exist between the study's definitions of adverse events and ClinicalTrials.gov definitions.
Arm/Group | Total Study Population
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
This study was conducted in healthy adult volunteers in a controlled laboratory environment, which may limit generalizability to clinical populations. The short intervention duration and immediate outcome assessments do not allow evaluation of longer-term effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT06228703/Prot_SAP_001.pdf